CLINICAL TRIAL: NCT00244686
Title: 104317: An Open-Label Compassionate Use Access and Long-Term Access Study of Anti IL-5 (Mepolizumab) Treatment in Subjects With Hypereosinophilic Syndrome. 201956: A Long-term Access Programme for Subjects With Severe Asthma Who Participated in a GSK-sponsored Mepolizumab Clinical Study. 112562: Expanded Access to Mepolizumab for Patients With Hypereosinophilic Syndrome
Brief Title: This Record Contains Information About the Mepolizumab Compassionate Use (CU) Product Activities: 104317: CU and Long-Term Access Study of Mepolizumab in HES. 201956:A Long-term Access Programme for Subjects With Severe Asthma 112562: Expanded Access for Patients With Hypereosinophilic
Status: No longer available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: MHE104317; 2007-000838-39 (EudraCT Number); NCT02543112 (obsolete NCT alias)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Hypereosinophilic Syndrome; Mepo; HES; Compassionate Use; Mepolizumab
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — mepolizumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Mepolizumab — open label investigational product

SUMMARY:
104317: The market authorisation application for mepolizumab for the indication of hypereosinophilic syndrome (HES) was filed in 2008, but later the file was withdrawn due to outstanding questions from regulator's raised from the application. On the basis of sponsor's evaluation, participants with life-threatening HES who have documented failure (lack of efficacy or a contra-indication) to at least 3 standard HES therapies (compassionate use) and participants who have participated in a previous GSK sponsored study in HES (long-term access) can be consider for mepolizumab treatment where the country regulation permits. In this study, participants will receive mepolizumab in an open-labelled manner, and limited data will be collected to evaluate the long-term safety and efficacy of mepolizumab.

201956: This is a Long-term Access Programme (LAP) which aims to support provision of mepolizumab, until it is commercially available, to eligible subjects with severe asthma who participated in a GSK-sponsored mepolizumab clinical study in severe asthma. Eligible subjects will initiate mepolizumab within a 6-month period following the individual subject's last scheduled visit in their preceding clinical study. For each subject benefit versus risk will be assessed throughout the study to support continued treatment with mepolizumab.

112562: To provide a mechanism for expanded access to mepolizumab therapy for eligible patients with HES. Whenever possible, use of an investigational medicinal product by a patient as part of a clinical trial is preferable. However, when patient enrollment in a clinical trial is not possible (such as when the patient is not eligible for ongoing clinical trials or the patient is not able to attend investigational sites), appropriate patients may receive mepolizumab through expanded access. This expanded access protocol was designed to allow access to mepolizumab for HES patients with seriously debilitating or life-threatening disease that are not able to enroll in clinical trials, including those patients that have already participated in a mepolizumab clinical trial.

ELIGIBILITY:
104317 Inclusion criteria:

* ≥ 12 years of age
* Has life-threatening HES as defined by the treating physician's documented view that likelihood of death is high unless the course of the disease is interrupted.
* Meets the diagnostic criteria for Hyper Eosinophilic Syndrome as defined by:

Eosinophilia >1500cells/ul for at least 6 months with evidence of symptoms and signs of organ system involvement or dysfunction that can be directly related to eosinophilia (with no evidence of parasitic, allergic or other recognized causes of eosinophilia such as connective tissues disease, malignancy) or Eosinophilia of >1500cells/ul for less than 6 months who meet the other criteria for HES accompanied by clear evidence of eosinophil tissue infiltration and with exclusion for secondary causes of eosinophilia as above.

* Compassionate use: Documented failure (lack of efficacy or a contra-indication) to at least 3 standard therapies (corticosteroids, cytotoxic agents, immunomodulatory therapy, and Imatinib mesylate) at the appropriate duration and dose
* Long-term access: Entry of subjects who participated in a previous GSK HES study to this study must be supported by the following: Subjects who received mepolizumab (if study treatment is known) in a previous GSK HES study: Documented improvement in symptoms and/or signs of HES following treatment with mepolizumab or Subjects who received mepolizumab or placebo in a previous GSK HES study: The treating physician must confirm a positive benefit/risk ratio, and the anticipated clinical benefit from mepolizumab must outweigh any potential safety or tolerability risk in this study or Subjects who participated in Study 200622 should complete the protocol required assessments for the duration of 32 weeks after randomization. Subsequently, subjects should complete the 20-week assessments in Study 205203, open-label extension (OLE) to Study 200622, prior to being considered for this protocol (MHE104317). In addition, subjects should not have had an adverse event (serious or non-serious) considered related to study treatment while participating in Study 200622 or Study 205203 which resulted in permanent withdrawal of study treatment.

104317 Exclusion Criteria:

* Subjects without HES but with other conditions associated with eosinophilic pathological process such as Churg-Strauss, Wegner's Granulomatosis, atopic disorders, hypersensitivity reactions to parasitic infections, eosinophilic gastroenteropathies, will not be eligible for this compassionate use program which is restricted to life-threatening HES.
* Female subjects of child -bearing potential who are not using an effective method of contraception:

Consistent and correct use of one of the following acceptable methods of birth control for one month prior to the start of the investigation product and 16 weeks after the last dose.

* Pregnant or lactating females
* Subjects with severe/life-threatening underlying disease unrelated to HES unrelated to HES where life expectancy is estimated to be less than 3 months.
* Subjects with a history of or current malignancy: Subjects with a history of or current lymphoma or Subjects with current malignancy or previous history of cancer in remission for less than 12 months prior to the first dose. Subjects that had localized carcinoma (i.e., basal or squamous cell) of the skin which was resected for cure will not be excluded.
* Subjects with history of serious allergic reaction (hypersensitivity/anaphylaxis) to anti-IL5 or other antibody therapy or known or suspected hypersensitivity to any component of mepolizumab, leading to treatment discontinuation
* Subjects with current drug or alcohol abuse where uncertain compliance with medication causes safety risk.
* subject currently receiving any other investigational product or other investigational intervention.

201956 Inclusion criteria:

* Subject participated in GSK-sponsored asthma clinical study with mepolizumab.
* Subject has either: completed the treatment period in the mepolizumab asthma clinical study to which they were originally enrolled or if the subject was withdrawn from study treatment prematurely during the mepolizumab asthma clinical study to which they were originally enrolled but the subject has completed the study assessments at the study visit that would have been the end of the respective treatment period.
* The treating physician requesting mepolizumab under this Long-term Access Programme considers the benefits of treatment with mepolizumab outweigh the risks for the individual subject.
* To be eligible for mepolizumab treatment under this Long-term Access Programme, females of childbearing potential (FCBP) must commit to consistent and correct use of an acceptable method of birth control, beginning with consent, for the duration of the treatment with mepolizumab and for 4 months after the last mepolizumab administration.
* The subject consents to receiving treatment with mepolizumab under this Long-term Access Programme. In the case of a paediatric subject being eligible a parent(s)/guardian will give written informed consent prior to the child's participation in the study. If applicable, the subject must be able and willing to give assent to take part in the study according to the local requirement.

201956 Exclusion criteria:

* A current malignancy or history of cancer in remission for less than 12 months (Subjects who had localized carcinoma (i.e., basal or squamous cell) of the skin which was resected for cure will not be excluded).
* Subject has other clinically significant medical conditions uncontrolled with standard-of-care therapy not associated with asthma, e.g., unstable liver disease, uncontrolled cardiovascular disease, ongoing active infectious disease requiring systemic treatment.
* Subject is pregnant or breastfeeding. Subjects should not be considered for continued treatment if they plan to become pregnant during the course of treatment with mepolizumab.
* Subject has a known allergy or intolerance to a monoclonal antibody or biologic therapy including mepolizumab.
* Subject had an adverse event (serious or non-serious) considered related to study treatment whilst participating in a clinical study with mepolizumab which resulted in permanent withdrawal of study treatment.
* Subject is receiving treatment with another biological therapy such as a monoclonal antibody therapy or intravenous (IV) immunoglobulin (Ig) therapy.
* Subjects who have received treatment with an investigational drug within the past 30 days or 5 terminal phase half-lives of the drug whichever is longer, prior to initiation of mepolizumab treatment under this Long-term Access Programme (this also includes investigational formulations of marketed products).
* Subject is currently participating in any other interventional clinical study.

112562 Inclusion criteria:

* In accordance with local procedures, written informed consent/assent can be obtained from the patient or legally authorized representative.
* ≥ 12 years of age at the time of signing the informed consent/assent.
* Meets the diagnostic criteria for HES as defined by:

Eosinophilia >1500 cells/µl for at least 6 months with evidence of symptoms and signs of organ system involvement or dysfunction that can be directly related to eosinophilia (with no evidence of parasitic, allergic or other recognised causes of eosinophilia such as connective tissues disease, malignancy) or Eosinophilia of >1500 cells/µl for less than 6 months and meet the other criteria for HES accompanied by clear evidence of eosinophil tissue infiltration and with exclusion of secondary causes of eosinophilia as above.

- Patients meeting all three of the following criteria will be eligible: The indication, HES, is a seriously debilitating or life-threatening disease; There is no satisfactory alternative treatment: documented failure (lack of efficacy or a contra-indication) to at least 3 standard therapies (corticosteroids, cytotoxic agents, immunomodulatory therapy, and Imatinib mesylate) at the appropriate duration and dose or demonstrated clinical benefit from prior treatment with mepolizumab; and There is reason to believe that the benefit:risk ratio for mepolizumab in the indication is positive.

112562 Exclusion criteria:

* Patients without HES but with other conditions associated with eosinophilic pathological processes such as eosinophilic granulomatosis with polyangiitis [EGPA], Wegener's granulomatosis, atopic disorders, parasitic infections, eosinophilic gastroenteropathies.
* Female patients of childbearing potential who are not using an effective method of contraception:

Consistent and correct use of an acceptable method of birth control for one month prior to the start of the investigational medicine and until 16 weeks after the last dose (see Appendix 3 for a list of acceptable methods of contraception).

* Pregnant or lactating females
* Patients with severe/life-threatening underlying disease unrelated to HES where life expectancy is estimated to be less than 3 months
* Patients with a history of or current malignancy:
* Patients with a history of or current lymphoma
* Patients with current malignancy or previous history of cancer in remission for less than 12 months prior to the first dose. Patients that had localized carcinoma (i.e., basal or squamous cell) of the skin which was resected for cure will not be excluded.
* Patients with history of serious allergic reaction (hypersensitivity/anaphylaxis) to anti-IL5 or other antibody therapy or known or suspected hypersensitivity to any component of mepolizumab, leading to treatment discontinuation
* Patients with current drug or alcohol abuse where uncertain compliance with the protocol and/or with the medical management instruction of the treating physician may cause safety risk
* Patients who have received treatment with an investigational agent (biologic or non-biologic, excluding mepolizumab) within the past 30 days or 5 drug half-lives whichever is longer, prior to the administration of mepolizumab under this protocol. The term "investigational" applies to any drug not approved for sale in the country in which it is being used or investigational formulations of marketed products.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Pavord I, Chan R, Brown N, Howarth P, Gilson M, Price RG, Maspero J. Long-term safety of mepolizumab for up to approximately 10 years in patients with severe asthma: open-label extension study. Ann Med. 2024 Dec;56(1):2417184. doi: 10.1080/07853890.2024.2417184. Epub 2024 Oct 28. PMID 39465531
- [Derived] Kuang FL, Fay MP, Ware J, Wetzler L, Holland-Thomas N, Brown T, Ortega H, Steinfeld J, Khoury P, Klion AD. Long-Term Clinical Outcomes of High-Dose Mepolizumab Treatment for Hypereosinophilic Syndrome. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1518-1527.e5. doi: 10.1016/j.jaip.2018.04.033. Epub 2018 May 8. PMID 29751154